CLINICAL TRIAL: NCT03388970
Title: Multicenter Randomized Controlled Trial of Vitamin K1 in the Treatment of Spontaneous Intracerebral Hemorrhage
Brief Title: Vitamin K1 in the Treatment of Spontaneous Intracerebral Hemorrhage
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HUANG XIANJIAN (Other)
Responsible Party: Sponsor-Investigator, HUANG XIANJIAN, vice professor, Shenzhen Second People's Hospital
Organization: Shenzhen Second People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUANGXIANJIAN20170608
Record Dates: First submitted 2017-10-29; First posted 2018-01-03 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Intracerebral Haemorrhage in Cerebellum
Keywords: vitamin K1; spontaneous intracerebral hemorrhage; effectiveness; outcome
MeSH Terms: interventions — Vitamin K 1; Saline Solution

STUDY DESIGN:
Masking Description: patient and family members
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- research group (Experimental): normal saline 100ml+ vitamin K1 20mg ivgtt qd day0 and day1。
  Interventions: Drug: Vitamin K 1
- placebo group (Placebo Comparator): normal saline100ml + normal saline 2 ml ivgtt qd day0 and day1
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Vitamin K 1 — Research group use Vitamin K1
  Arms: research group
Drug: normal saline — Placebo group use normal saline
  Arms: placebo group

SUMMARY:
In order to determine the effectiveness and safety of early vitamin K1 use in reducing the risk of bleeding and improving prognosis in patients with spontaneous intracerebral hemorrhage. Patients with spontaneous intracerebral hemorrhage (excluding rupture of aneurysm and vascular malformation) will be randomly divided into experimental group and control group. All the patients in the two groups were treated according to the guideline of spontaneous intracerebral hemorrhage. Patients in the experimental group was treated with intravenous injection of vitamin K1 20mg once a day for 2 days after admission, and the patients in control group was treated with normal saline as a control. The hematoma volume, coagulation function, platelet levels and GCS scales of the two groups will be recorded in 0d, 1d, 3d, 7d post bleeding stroke, furthermore, length of ICU stay and total hospitalization, incidence of complications during hospitalization are to be recorded. During the follow-up, mRS score will be recorded at 1m and 6m post bleeding stroke.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage is a common disease in the department of neurosurgery, which often leads to long-term coma and severe neurological dysfunction. The amount of cerebral hemorrhage is directly related to the prognosis of the patients, and a small number of patients still suffer from the adverse consequences of delayed bleeding after active treatment. Vitamin K1 is a necessary ingredient in the liver to produce clotting factors II, VII, IX, and X, and vitamin K1 supplementation increases clotting function. On the contrary, vitamin K1 increases the risk of thrombosis. In this study, patients with spontaneous intracerebral hemorrhage (excluding rupture of aneurysm and vascular malformation) will be randomly divided into experimental group and control group. All the patients in the two groups were treated according to the guideline of spontaneous intracerebral hemorrhage. Patients in the experimental group was treated with intravenous injection of vitamin K1 20mg once a day for 2 days after admission, and the patients in control group was treated with normal saline as a control. The hematoma volume, coagulation function, platelet levels and GCS scales of the two groups will be recorded in 0d, 1d, 3d, 7d post bleeding stroke, furthermore, length of ICU stay and total hospitalization, incidence of complications during hospitalization are to be recorded. During the follow-up, mRS score will be recorded at 1m and 6m post bleeding stroke. Finally, the effectiveness and safety of early vitamin K1 use in reducing the risk of bleeding and improving prognosis in patients with spontaneous intracerebral hemorrhage will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracerebral hemorrhage (Non - aneurysmal or arteriovenous malformations which confirmed by cerebral arterial CT enhancement or DSA);
* Age 18-65 years, male or non-pregnant female;
* GCS score at admission (4 to12);
* during the hospitalization, no urokinase and other hemostatic drugs were used except for etamsylate and vitamin K1;
* informed consent signed by the patient's family

Exclusion Criteria:

* irregular lobulated hematoma (volume of hematoma can not be calculated accurately), such as intraventricular hemorrhage;
* severe liver disease or impaired liver function;
* pregnant or lactating women;
* history of using anticoagulation or antiplatelet aggregation drug (including Cilostazol, aspirin, dipyridamole, heparin, low molecular weight heparin, hirudin, dabigatran, and warfarin);
* non-accepted informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
The volume of cerebral hemorrhage | Day0
  The volume of cerebral hemorrhage at certain time post onset（ml）
The volume of cerebral hemorrhage | Day3
  The volume of cerebral hemorrhage at certain time post onset（ml）
The volume of cerebral hemorrhage | Day7
  The volume of cerebral hemorrhage at certain time post onset（ml）

SECONDARY OUTCOMES:
The Activated Partial Thromboplastin Time（s）at certain time post onset | Day0
  Activated Partial Thromboplastin Time（s）
The Activated Partial Thromboplastin Time（s）at certain time post onset | Day3
  Activated Partial Thromboplastin Time（s）
The Activated Partial Thromboplastin Time（s）at certain time post onset | Day7
  Activated Partial Thromboplastin Time（s）
The condition of Platelet level at certain time post onset | Day0
  The condition of Platelet level at certain time post onset（10^9/L）
The condition of Platelet level at certain time post onset | Day3
  The condition of Platelet level at certain time post onset（10^9/L）
The condition of Platelet level at certain time post onset | Day7
  The condition of Platelet level at certain time post onset（10^9/L）
The condition of GCS scale post(3-15) at certain time post onset | Day0
  The condition of GCS scale post(3-15) at certain time post onset
The condition of GCS scale post(3-15) at certain time post onset | Day3
  The condition of GCS scale post(3-15) at certain time post onset
The condition of GCS scale post(3-15) at certain time post onset | Day7
  The condition of GCS scale post(3-15) at certain time post onset
The prothrombin time(s) at certain time post onset | Day0
  prothrombin time(s)
The prothrombin time(s) at certain time post onset | Day3
  prothrombin time(s)
The prothrombin time(s) at certain time post onset | Day7
  prothrombin time(s)
The Fibrinogen (g/L)at certain time post onset | Day0
  Fibrinogen (g/L)
The Fibrinogen (g/L)at certain time post onset | Day3
  Fibrinogen (g/L)
The Fibrinogen (g/L)at certain time post onset | Day7
  Fibrinogen (g/L)
The Thrombin Time(s) at certain time post onset | Day0
  Thrombin Time(s)
The Thrombin Time(s) at certain time post onset | Day3
  Thrombin Time(s)
The Thrombin Time(s) at certain time post onset | Day7
  Thrombin Time(s)

OTHER OUTCOMES:
length of stay in ICU | about two weeks
  length of stay in ICU
Total hospital stay | about one month
  Total hospital stay
Complications1 | 6 month post onset
  neurologic complications
The Modified Rankin Scale (mRS) | month 1 post onset
  The scale runs from 0-6, running from perfect health without symptoms to death.0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6 - Dead.
The Modified Rankin Scale (mRS) | month 6 post onset
  The scale runs from 0-6, running from perfect health without symptoms to death.0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6 - Dead.
Complications2 | 6 month post onset
  infection complications
Complications3 | 6 month post onset
  complications of coagulation

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Shenzhen second people's hospital, Shenzhen, Guangdong
  - The fifth people's hospital of Longgang District, Shenzhen, Shenzhen, Guangdong
  - Baoan District central hospital of Shenzhen, Shenzhen, Guangdong
  - Shajing hospital of Baoan District ,Shenzhen, Shenzhen, Guangdong
  - The second People's hospital of Longgang District, Shenzhen, Shenzhen, Guangdong

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-10-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03388970/SAP_000.pdf
  • Informed Consent Form (2017-10-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03388970/ICF_001.pdf
  • Study Protocol (2017-10-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03388970/Prot_002.pdf